CLINICAL TRIAL: NCT05038514
Title: The Effect of Music Therapy on Adaptation and Anxiety Levels in COVID-19 Patients Given Prone Position: A Triple-blind Randomized Controlled Clinical Trial
Brief Title: The Effect of Music Therapy in COVID-19 Patients Given Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Senay Takmak, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2100014997
Record Dates: First submitted 2021-09-05; First posted 2021-09-09 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Music Therapy; Anxiety; Respiratory Distress Syndrome; Intensive Care Units; Nursing
Keywords: COVID-19; Prone position
MeSH Terms: conditions — Anxiety Disorders; Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: A triple-blind randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind (i.e., triple-masking) studies are randomized experiments in which the treatment or intervention is unknown to (a) the research participant, (b) the individual(s) who administer the treatment or intervention, and (c) the individual(s) who assess the outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy (Experimental): Music therapy intervention, bluetooth headphones will be applied in the intensive care unit and will be disinfected after the application. The intervention consists of a 30-minute, single-session, nature-based music concert. the music concert is calibrated by the audiologist (60 decibels). During nature-based music listening, patients will be asked to close their eyes, rest and follow the sound flow.
  Interventions: Other: musıc therapy
- control (No Intervention): The control group will be given the prone position and music therapy will not be applied.

INTERVENTIONS:
Other: musıc therapy — After the prone position was given to the patients, according to the randomization table, the intervention group was given 30 minutes by the nurse. nature-based music therapy will be applied.
  Arms: music therapy

SUMMARY:
Almost half of the patients diagnosed with COVID-19 pneumonia develop ARDS and most of these patients are treated in the intensive care unit. In the management of COVID-19 ARDS, prone position is applied to improve physiological parameters by facilitating better distribution of tidal volume and drainage of secretions. It has been reported that awake patients in COVID clinics could not adapt their prone position due to anxiety . Jiang et al (2020) reported that awake patients may not tolerate the prone position and may experience anxiety due to posture habits and discomfort.

It was determined that anxiety developed on the second day of hospitalization in the intensive care unit, state anxiety was associated with trait anxiety and pain, and anxiety was low in patients receiving mental health care/treatment . And also not to change position himself of patient in prone position due to care equipment etc it can cause loss of self-control and anxiety. Twelve-sixteen hour prone position recommendation for clinical improvement, positioning difficulties in patients who cannot position themselves may also trigger anxiety in awake patients It has been suggested that music therapy may be effective in reducing anxiety related to weaning from mechanical ventilation in COVID-19 patients. Music therapy intervention in ICU has been tested in sessions of at least 30 minutes, 1-30 days, with options such as western music, classical Chinese music, nature-based music. In the study of Chu and Zhang (2021), it was shown that the recovery time for tomography findings, the number of days of hospital stay and the rates of transfer to the intensive care unit were lower in the patient group who received holistic mode including traditional Chinese medicine, music therapy, and emotional support in COVID-19 patients. Studies evaluating the effectiveness of music therapy alone in the COVID-19 intensive care process could not be reached. It is thought that music therapy applied in the prone position in the COVID-19 intensive care unit will reduce the anxiety of the patients, adapt to the prone position and improve their clinical parameters.

DETAILED DESCRIPTION:
The Corona virus disease 2019 Pandemic (COVID-19) has caused a psychosocial depression in the world. Acute severe or critical condition has been observed in 20% of individuals diagnosed with COVID-19. It is stated that viral pneumonia or Acute Respiratory Distress Syndrome (ARDS) and organ failures develop in these individuals. Almost half of the patients diagnosed with COVID-19 pneumonia develop ARDS and most of these patients are treated in the intensive care unit. In the management of COVID-19 ARDS, prone position is applied to improve physiological parameters by facilitating better distribution of tidal volume and drainage of secretions. It is thought that the prone position will be more effective in the early stages of the disease and awake patients. It is recommended that the prone position especially in moderate to severe ARDS cases be applied for at least 12 hours after symptoms stabilize. Elkattawy and Noori (2020) reported that at least 6-8 hours of prone position improves oxygenation in the COVID-19 case without ARDS criteria. Mac Sweeney et al. (2020) reported that clinical parameters improved, intubation and ventilator requirement were delayed in an awake, self-prone COVID-19 case. However, Somagutta et al (2021) reported anxiety, back pain, adjustment and tolerance problems in awake and not mechanically ventilated patients. Bastoni et al, in the study which they evaluated prone adapt at emergency department in Italy; it is reported positioning could not be maintained in four out of ten patients due to unconformity, pain, and rejection of prone position. It has been reported that awake patients in COVID clinics could not adapt their prone position due to anxiety. Jiang et al (2020) reported that awake patients may not tolerate the prone position and may experience anxiety due to posture habits and discomfort.

It was determined that anxiety developed on the second day of hospitalization in the intensive care unit, state anxiety was associated with trait anxiety and pain, and anxiety was low in patients receiving mental health care/treatment. And also not to change position himself of patient in prone position due to care equipment etc it can cause loss of self-control and anxiety. Twelve-sixteen hour prone position recommendation for clinical improvement, positioning difficulties in patients who cannot position themselves may also trigger anxiety in awake patients.

Music therapy is applied as a non-pharmacological nursing intervention in the anxiety management of patients in intensive careIt is stated that music therapy is effective in stress-anxiety management, improves vital signs and sleep quality, and may have a muscle relaxant effect in interventions applied in covid-19. It has been suggested that music therapy may be effective in reducing anxiety related to weaning from mechanical ventilation in COVID-19 patients. Music therapy intervention in ICU has been tested in sessions of at least 30 minutes, 1-30 days, with options such as western music, classical Chinese music, nature-based music. It has been reported that music therapy applied with all types of music provides normal heart rate, respiratory recovery and muscle relaxation. Golino et al. listened to music for 30 minutes according to the preferences of the patients in the intensive care unit and their vital signs, pain and anxiety were evaluated. While there was an improvement in heart rate and respiration, oxygen saturations did not change. At the same time, patients reported less pain and anxiety. In the study of Chu and Zhang (2021), it was shown that the recovery time for tomography findings, the number of days of hospital stay and the rates of transfer to the intensive care unit were lower in the patient group who received holistic mode including traditional Chinese medicine, music therapy, and emotional support in COVID-19 patients. Studies evaluating the effectiveness of music therapy alone in the COVID-19 intensive care process could not be reached. It is thought that music therapy applied in the prone position in the COVID-19 intensive care unit will reduce the anxiety of the patients, adapt to the prone position and improve their clinical parameters.

Objective: The aim of this study is to evaluate the effect of music therapy applied in the prone position on anxiety, compliance with the prone position, and vital signs in patients diagnosed with COVID-19 in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18-80
* Developing respiratory failure due to COVID-19
* Prone position applied
* Staying in intensive care unit for at least 24 hours
* Awake and cooperative
* Recipient of oxygen mask or high-flow oxygen therapy or noninvasive mechanical ventilation support
* Stable hemodynamic status

Exclusion Criteria:

* Those who do not agree to participate in the research
* Those with communication barrier problems
* Intubated
* Sedation drug applied
* Those who need emergency intervention during work
* Having a diagnosis of neurological and psychological medicine
* Abnormal deterioration in physiological parameters
* Patients transferred to another service or discharged
* patients with hearing impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
anxiety | change from baseline state anxiety after position change at one day
  State Anxiety Inventory
vital signs | change from baseline pulse rate after position change at one day
  pulse rate
vital signs | change from baseline respiratory rate after position change at one day
  respiratory rate
vital signs | change from baseline blood pressure after position change at one day
  blood pressure
vital signs | change from baseline oxygen saturation after position change at one day
  oxygen saturation
prone position adaptation | time/hour to stay in prone position at one day
  length of stay in prone position

CONTACTS AND LOCATIONS:
Overall Officials: Halil İbrahim KARAÇAR, RN, Study Chair — Antalya Kepez State Hospital Intensive Care Unit
Locations (1):
- Antalya Kepez State Hospital Intensive Care Unit, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The decision to share the study results will be made during the study period or when it is concluded.

REFERENCES:
- [Background] Bamford, P., Bentley, A., Dean, J., Whitmore, D. & Wilson-Baig, N. ICS guidance for prone positioning of the conscious COVİD-19 patient 2020. London: Intensive Care Society, 2020. (01.10.2020 tarihinde https://emcrit.org/wp-content/uploads/2020/04/2020-04-12-Guidance-for-conscious-proning.pdf adresinden ulaşılmıştır).
- [Background] Bastoni D, Poggiali E, Vercelli A, Demichele E, Tinelli V, Iannicelli T, Magnacavallo A. Prone positioning in patients treated with non-invasive ventilation for COVID-19 pneumonia in an Italian emergency department. Emerg Med J. 2020 Sep;37(9):565-566. doi: 10.1136/emermed-2020-209744. Epub 2020 Jul 6. PMID 32748797
- [Background] Chu L, Zhang Y. A study on nursing effect of integrated traditional Chinese and Western medicine management mode on COVID-19. Jpn J Nurs Sci. 2021 Mar 7;18(3):e12411. doi: 10.1111/jjns.12411. Online ahead of print. PMID 33682284
- [Background] Dwitasari, M. A. D., & Laksmidewi, A. A. A. P. (2020). Convalescent Plasma Therapy in Effort of Weaning from Mechanical Ventilation Using Music Stimulation in Severe COVİD-19 Patients. Open Access Macedonian Journal of Medical Sciences, 8(T1), 192-197.
- [Background] Elkattawy S, Noori M. A case of improved oxygenation in SARS-CoV-2 positive patient on nasal cannula undergoing prone positioning. Respir Med Case Rep. 2020 May 4;30:101070. doi: 10.1016/j.rmcr.2020.101070. eCollection 2020. PMID 32368483
- [Background] Gibson PG, Qin L, Puah SH. COVID-19 acute respiratory distress syndrome (ARDS): clinical features and differences from typical pre-COVID-19 ARDS. Med J Aust. 2020 Jul;213(2):54-56.e1. doi: 10.5694/mja2.50674. Epub 2020 Jun 22. No abstract available. PMID 32572965
- [Background] Golino AJ, Leone R, Gollenberg A, Christopher C, Stanger D, Davis TM, Meadows A, Zhang Z, Friesen MA. Impact of an Active Music Therapy Intervention on Intensive Care Patients. Am J Crit Care. 2019 Jan;28(1):48-55. doi: 10.4037/ajcc2019792. PMID 30600227
- [Background] Hunter BC, Oliva R, Sahler OJ, Gaisser D, Salipante DM, Arezina CH. Music therapy as an adjunctive treatment in the management of stress for patients being weaned from mechanical ventilation. J Music Ther. 2010 Fall;47(3):198-219. doi: 10.1093/jmt/47.3.198. PMID 21275332
- [Background] Latuapo, A., Farid, M., & Ab Rahman, Z. (2020). Pharmaceutıcal and Nonpharmaceutıcal Use Of Musıc and Al-Quran Therapy in Preventıng The Spread Of Pandemıcs (Covıd-19): A Systematıc Revıew. Systematic Reviews in Pharmacy, 11(12), 1171-1179.
- [Background] Shang Y, Pan C, Yang X, Zhong M, Shang X, Wu Z, Yu Z, Zhang W, Zhong Q, Zheng X, Sang L, Jiang L, Zhang J, Xiong W, Liu J, Chen D. Management of critically ill patients with COVID-19 in ICU: statement from front-line intensive care experts in Wuhan, China. Ann Intensive Care. 2020 Jun 6;10(1):73. doi: 10.1186/s13613-020-00689-1. PMID 32506258
- [Background] Somagutta, M. R., Pormento, M. K. L., Khan, M. A., Hamdan, A., & Dodla, S. N. (2021). 262: Awake Self Prone Positioning Outcomes in Nonintubated COVİD-19 Patients. Critical Care Medicine, 49(1), 118.
- [Background] Wormser J, Romanet C, Philippart F. Prone position in wards for spontaneous breathing Covid-19 patients: a retrospective study. Ir J Med Sci. 2021 Nov;190(4):1519-1522. doi: 10.1007/s11845-020-02479-x. Epub 2021 Jan 15. PMID 33449332
- [Background] Froutan R, Eghbali M, Hoseini SH, Mazloom SR, Yekaninejad MS, Boostani R. The effect of music therapy on physiological parameters of patients with traumatic brain injury: A triple-blind randomized controlled clinical trial. Complement Ther Clin Pract. 2020 Aug;40:101216. doi: 10.1016/j.ctcp.2020.101216. Epub 2020 Jun 30. PMID 32891292